CLINICAL TRIAL: NCT05118308
Title: Endoscopic Ultrasound Guided Liver Biopsy and Portal Pressure Gradient Measurement Compared to the Transjugular Approach: a Randomized Controlled Trial
Brief Title: EUS vs TJ for Liver Biopsy and Portal Pressure Gradient Measurement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Amine Benmassaoud, Principal investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2021.7601
Record Dates: First submitted 2021-10-22; First posted 2021-11-11 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Portal Hypertension; Chronic Liver Disease; Cirrhosis
Keywords: eus-portal pressure gradient; eus-liver biopsies; liver biopsy; portal pressure gradient; hepatic venous pressure gradient; transjugular-portal pressure gradient; Transjugular-Liver biopsies
MeSH Terms: conditions — Hypertension, Portal; Fibrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: As EUS and TJ procedures are inherently different, patients and health-care workers directly involved in the procedure, including nurses, physicians, and technicians, will not be blinded. Pathologists interpreting liver biopsies will be blinded to the intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Transjugular approach (Experimental): Transjugular hepatic venous pressure gradient measurement with liver biopsy (HVPG-LB).
  Interventions: Procedure: Transjugular hepatic venous pressure gradient measurement with liver biopsy
- Endoscopic ultrasound approach (Experimental): Endoscopic ultrasound portal pressure gradient measurement with liver biopsy (EUS-PPG-LB)
  Interventions: Procedure: Endoscopic ultrasound portal pressure gradient measurement with liver biopsy

INTERVENTIONS:
Procedure: Transjugular hepatic venous pressure gradient measurement with liver biopsy — This procedure will be performed by an experienced interventional radiologist who will be supported by a radiology technician and nurse. Transjugular hepatic venous pressure gradient measurement will be performed using standard procedure. Following this, a transjugular liver biopsy will be obtained using an 18-gauge transjugular liver biopsy needle.
  Arms: Transjugular approach
Procedure: Endoscopic ultrasound portal pressure gradient measurement with liver biopsy — A linear echoendoscope is inserted with the patient under conscious sedation. Using a through the scope 25-gauge needle connected to a digital manometer, portal and hepatic veins will be punctured under EUS guidance from a trans-gastric/hepatic approach. Following this, EUS-Liver biopsy is then performed immediately following EUS-PPG using a 19-gauge fine needle biopsy (FNB).
  Arms: Endoscopic ultrasound approach

SUMMARY:
This study will directly compare the endoscopic ultrasound guided approach to obtain adequate liver biopsies and portal pressure gradient measurements to the current standard of care which uses the transjugular approach.

DETAILED DESCRIPTION:
Current guidelines recommend that when a hepatic venous pressure gradient and a liver biopsy are needed, the liver biopsy should be done by the transjugular approach during the same session. A major limitation is that liver biopsies obtained by the transjugular approach meet quality criteria proposed by the American Association for the Study of Liver Diseases (at least 2-3cm with at least 11 complete portal tracts) in only 40% of cases.

Recent studies have shown that endoscopic ultrasound-guided liver biopsy (EUS-LB) can achieve a high rate of adequate liver biopsies using the same strict criteria described above. In addition, a novel endoscopic-ultrasound adapted manometer allows the safe and accurate measurement of portal pressure gradient (PPG) which correlates well with hepatic venous pressures (HVPG) obtained by the transjugular approach. Unfortunately to this day, no randomized controlled trials has compared the EUS-LB and PPG vs TJ-LB and HVPG directly.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Undergoing evaluation for chronic liver disease or portal hypertension
* Planned to undergo a liver biopsy and HVPG by their treating hepatologist for clinical purposes
* Signed informed consent

Exclusion Criteria:

* Uncorrectable coagulopathy (INR above 1.5)
* Uncorrectable thrombocytopenia (Platelets under 50,000)
* Anticoagulation or antiplatelet therapy that cannot be discontinued
* Surgically altered upper digestive anatomy
* Biliary obstruction
* Grade II ascites or more
* Intrahepatic portal vein thrombosis
* Previous liver transplantation
* Past hypersensitivity reaction to midazolam or ketamine
* History of psychotic disorder
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Compare the proportion of adequate Liver Biopsy specimens with reliable portal pressure gradient obtained by TJ or EUS | 2 weeks
  Liver Biopsy (LB) specimens are defined as a biopsy of at least 25mm in length following formalin fixation and at least 11 complete portal tracts. The Portal pressure gradient (PPG) measurement is defined as two PPG values with less than 2mmHg difference.

SECONDARY OUTCOMES:
Technical success | 1 day
  Compare the proportion of HVPG and LB obtained by TJ or EUS approach
Liver biopsy-related outcomes | 2 weeks
  Number of adequate liver biopsies obtained, total aggregate length (defined as the sum of the lengths of all specimens following fixation), number of complete portal tracts per specimen, and total number of passes needed.
PPG-related outcomes | 1 day
  Number of PPG obtained, number of reliable PPG obtained
Adverse events | 30 days
  Proportion of adverse events in the TJ and EUS arms following the procedure, at day 7, and day 30.
Satisfaction with sedation | 1 day
  Compare the score obtained on the sedation satisfaction surveys as completed by the participant and the physician within the 2 arms

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benmassaoud A, Bessissow A, Samoukovic G, Wong P, Zhao X, Deschenes M, Sebastiani G, Cabrera T, Valenti D, Boucher LM, Pelage JP, Muchantef K, Cardenas A, Givis MA, White S, Bousquet-Dion G, Waked C, Jacques J, Rahme E, Geraci O, Martel M, Barkun A, Maedler-Kron C, Chen YI. EUS-Guided Liver Biopsy and Portal Pressure Measurement Compared With a Transjugular Approach: A Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2025 Oct 3:S1542-3565(25)00850-X. doi: 10.1016/j.cgh.2025.09.025. Online ahead of print. PMID 41046961